CLINICAL TRIAL: NCT00377689
Title: Evaluation of an Intervention Program Targeted at Improving Balance and Functional Skills After Stroke - a Randomized Controlled Study
Brief Title: Evaluation of an Intervention Program Targeted at Improving Balance and Functional Skills After Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Vardalinstitutet The Swedish Institute for Health Sciences (Other); Erik & AnnMarie Detlofs Foundation (Unknown); The Swedish National Stroke society (Unknown); The Northern County Councils Regional Federation (Unknown)
Responsible Party: Umea University, Mrs Eva Holmgren, RPt, PhD student, Umea University
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: Dnr 04-022
Record Dates: First submitted 2006-09-15; First posted 2006-09-18 (Estimated); Last update posted 2008-10-29 (Estimated); Status verified 2008-10

CONDITIONS: Cerebrovascular Accident; Musculoskeletal Equilibrium
Keywords: Accidental falls; Cerebrovascular accident; Balance; ADL; Self efficacy; Quality of Life; Gait parameters
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

INTERVENTIONS:
Behavioral: high intensity functional exercise — high intensity functional exercise

SUMMARY:
The purpose of this study is to evaluate a 5-week intervention program targeted at improving balance and functional skills for people with stroke.

DETAILED DESCRIPTION:
Many people with stroke experience a deterioration in balance and a functional decline due to hemiplegic muscle strength. This tend to restrict the persons activity in daily life and also leads to a low falls self efficacy.

High intensity exercise have shown to be effective for improving strength and balance for older people in general living in residential care facilities. It is interesting to see if this high intensity exercise also is applicable in the older stroke population.

Comparison: An intervention group receives three training sessions per week and one theory session per week during 5 weeks, compared to a control group that receives one theory session per week during 5 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 55 years of age or older
* stroke diagnosis 3-6 months prior to inclusion
* ability to walk 10 meter with or without assistive device
* ability to understand simple instructions

Exclusion Criteria:

* TIA
* independent in walking outdoors
* serious visual impairment
* serious hearing impairment
* long distance to intervention station

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2006-09; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Improvement in balance | post, 3 & 6 months

SECONDARY OUTCOMES:
Reduced falls | post, 3 & 6 months
Improved self-efficacy | post, 3 & 6 months
Improved ADL | post, 3 & 6 months
Improved walking ability | post, 3 & 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Eva Holmgren, PhD student, Principal Investigator — Umeå University & The Vårdal Institute; Per Wester, MD Professor, Study Chair — Umeå University
Locations (1):
- Umeå University, department of Community science and rehabilitation, Umeå, Sweden